CLINICAL TRIAL: NCT03549949
Title: Nationwide Awareness Campaign and Call for Dental Screening for HHT in Germany
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Essen (Other)
Collaborators: Philipps University Marburg (Other); University Hospital, Aachen (Other); German HHT self-help group (Unknown)
Responsible Party: Principal Investigator, Urban Geisthoff, Prof. Dr. med., Philipps University Marburg
Other Study IDs: Dental Screening for HHT
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Dental Diseases
Keywords: pulmonary arteriovenous malformations
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Stomatognathic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HHT is a relative rare autosomal dominant inherited disorder of the fibrovascular tissue. Diagnosis of HHT is often delayed for decades (Pierucci 2012). However, it would be desirable to achieve an early diagnosis as early screening and treatment decrease disease-associated complications and increase life expectancy (Kroon 2018). Our approach is a nationwide call and awareness campaign to dentists in Germany, as nearly all persons visit a dentist from time to time. This approach is promising to us, as most patients develop nosebleeds and multiple, typical telangiectases of the skin or mucosa. A predilection site is the oral mucosa and the face, including the lips (Shovlin 2000).

DETAILED DESCRIPTION:
The German self-help group is taking down the number of inquiries from patients and physicians per months since April 2017. In June 2018 an article about HHT is planned to be published in the journal of the German dental association and the Federal Association of Fund Dentists of Germany. This journal is distributed to all dentists in Germany and is a set book for them. Total circulation in 2017 was 77,621 (http://www.aerzteverlag.de/portfolio/fachwissen-medizindental/zm-zahnaerztliche-mitteilungen/profil/ ). The article describes the case of visceral abscesses after dental screening in a patient with HHT and pulmonary arteriovenous malformations. These could probably have been prevented if the dentist had prescribed an antibiotic prophylaxis to the patient. The article includes a call to search for telangiectases. If those are seen the dentist is recommended to ask the patient if he or relatives have nosebleeds. If both apply, the dentist is asked to inform the patient about HHT and give him the address of the national German self-help group.

After 3 and 6 months a reminder shall be published in the same journal.

ELIGIBILITY:
Inclusion Criteria:

* patients having telangiectasia and nosebleeds or nosebleeds in the family

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Telagiectases seen by the dentist should lead to the question if the patient or relatives have nosebleeds. If both apply, the dentist is asked to inform the patient about Hereditary Hemorrhagic Telangiectasia and give the address of the national German self-help group to the patient.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of inquiries to the German self-help group | 1 year
  Number of inquiries to the German self-help group before and after publication of the articles.

SECONDARY OUTCOMES:
Number of specific HHT diagnosis in the information system for health services (Informationssystem Versorgungsforschung) of the national German institute for medical documentation and information (DIMDI) | 1 year
  The number of specific HHT diagnosis in the information system for health services (Informationssystem Versorgungsforschung) of the national German institute for medical documentation and information (DIMDI) will be analyzed for potential changes.

CONTACTS AND LOCATIONS:
Overall Officials: Urban Geisthoff, Prof. Dr. med., Principal Investigator — Philipps University Marburg
Locations (1):
- University Hospital Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shovlin CL, Guttmacher AE, Buscarini E, Faughnan ME, Hyland RH, Westermann CJ, Kjeldsen AD, Plauchu H. Diagnostic criteria for hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber syndrome). Am J Med Genet. 2000 Mar 6;91(1):66-7. doi: 10.1002/(sici)1096-8628(20000306)91:13.0.co;2-p. PMID 10751092
- [Background] Pierucci P, Lenato GM, Suppressa P, Lastella P, Triggiani V, Valerio R, Comelli M, Salvante D, Stella A, Resta N, Logroscino G, Resta F, Sabba C. A long diagnostic delay in patients with Hereditary Haemorrhagic Telangiectasia: a questionnaire-based retrospective study. Orphanet J Rare Dis. 2012 Jun 7;7:33. doi: 10.1186/1750-1172-7-33. PMID 22676497
- [Background] Kroon S, Snijder RJ, Faughnan ME, Mager HJ. Systematic screening in hereditary hemorrhagic telangiectasia: a review. Curr Opin Pulm Med. 2018 May;24(3):260-268. doi: 10.1097/MCP.0000000000000472. PMID 29470256